CLINICAL TRIAL: NCT05157139
Title: Clinical Trial for Oral Formula of Vanillin and Wheat Germ Oil for Treatment of Mild and Moderate COVID-19 Viral Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Collaborators: Assoc. Prof. Ayman Ibrahim Baess (Unknown); Dr. Noha Alaa Eldine Hassan Hamdy (Unknown); Ph. Hanya Hesham Sweilam (Unknown)
Responsible Party: Principal Investigator, Ahmed Ibrahim ElMallah, Professor of Pharmacology & Therapeutics, Faculty of Pharmacy, Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0106922
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-12

CONDITIONS: Mild-to-moderate COVID-19
Keywords: mild-to-moderate COVID-19 vanillin, wheat germ oil
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients receiving only standard care
- Intervention (low dose) (Active Comparator): Two capsules twice daily for 3 days then one capsule twice daily for 2 days
  Interventions: Drug: Oral Capsule
- Intervention (high dose) (Active Comparator): two capsules three times daily for 3 days, followed by one capsule three times daily for 4 days
  Interventions: Drug: Oral Capsule

INTERVENTIONS:
Drug: Oral Capsule — Oral Capsule of vanillin & wheat germ oil
  Arms: Intervention (high dose); Intervention (low dose)

SUMMARY:
* The study is a randomized clinical trial to assess a natural formula of vanillin & wheat germ oil to treat and stop the clinical progression of COVID-19.
* The study aims to treat people with mild-to-moderate COVID-19 before their cases become severe.
* The study duration is a 5-day experimental intervention and an extended 4 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

1. PCR confirmed diagnosis for COVID-19.
2. Age ≥18 years.
3. Both genders
4. The disease started within 7 days (ideally 72 hours) of diagnosis or clinical deterioration.
5. Patients diagnosed as mild or moderate

Exclusion Criteria:

1. Patients diagnosed with severe Illness: Individuals who have SpO2 <92% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, respiratory frequency >30 breaths/min, or lung infiltrates >50%.
2. General: advanced kidney disease; advanced liver disease; pregnancy (known or potential) or lactation, and advanced cardiovascular diseases.
3. Allergy to Vanilla flavor, vanillin, or wheat germ oil
4. Active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
1. Mean change in the disease severity (clinical assessment). | 3-5 days
  Time taken for the changes from moderate or mild or complete recovery/FDA assessment of key COVID-19-related symptoms score
2. Rate of disease remission. | 3-5 days
  For mild/moderate symptoms patients: fever, cough and other symptoms relieved
3. Hospitaization & Survival rate | up to 4 weeks
  Comparing the influence of the intervention on the hospitalization & Survival rate followed for up to 4 weeks.

SECONDARY OUTCOMES:
4. Mean change in complete blood picture | 3-5 days
  CBC
5. Mean change in C reactive protein (CRP) | 3-5 days
  CRP
9. The mean change in serum interleukin-6 (IL-6) | 3-5 days
  serum IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The research team will share after results
Time Frame: up to March 2022